CLINICAL TRIAL: NCT03700463
Title: Assessment of Executive Functions in Preterm Children in 3 to 4 Year Old From Behavioral Rating Inventory of Executive Function (BRIEF) Questionnaire
Brief Title: Executive Functions and Preterm Children in 3 to 4 Year Old
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC18_0147
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Preterm Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: BRIEF parental survey — Estimate incidence of executive functions disorders in preterm children in 3 to 4 year old, born less than 34 weeks of gestation

SUMMARY:
Preterm children have a high risk for neurodevelopmental impairments. The impact on motor functions and neurosensory functions is demonstrated but the incidenceof executive functions is not described for preterm infants.

DETAILED DESCRIPTION:
It is an epidemiologic, observational, prospective study. All patients, included in the LIFT cohort, in 3 to 4 year old during the period study, are contacted by mail. Patientswith congenital anomalies or genetic syndromes are excluded. Children with parents who do not speak French are excluded. Antenatal and postnatal criteria known to be associated with disorders of executive functions are collected as, gestational age, sex, multiple pregnancy, intrauterine growth retardation, antenatal or postnatal steroid use, breastfeeding, cerebral injuries and socio-economic status. After a couple of weeks, parents are contacted by a study manager, by phone call, to collect parental consent and answer parental questions. After consent collect, BRIEF questionnaires are sending. If they wish, parents could give the BRIEF teacher questionnaire to the mean teacher. Teachers send by themselves their response. An informatic version is available with a personal link given especially by mail for each child. All data are anonymous. BRIEF questionnaire is composed of 63 items, exploring 2 main domains: behavior and metacognition. Twenty minutes are necessary to complete questionnaire. In case of no questionnaire return after one month, parents are contacted by phone. The investigators hypothesize a lost to follow-up at 0.25 and no response at 0.35. The response expected is 300 questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* patient in 3 to 4 year old, included in LIFT cohort

Exclusion Criteria:

* Congenital abnormalities including nervous system malformations; genetic diseases; incomplete understanding of written and oral French by parents

Ages: 3 Years to 4 Years | Sex: All
Age Groups: Child
Study Population: patients which former preterm of gestational age less than 34 weeks
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence of disorders of executive functions in 3 to 4 year old which former preterm of gestational age less than 34 weeks, from the Behavioral Rating Inventory of Executive Function questionnaire. | 3 to 4 years after preterm birth
  sum of 63 items is calculated

SECONDARY OUTCOMES:
neonatal factors | 3 to 4 years after preterm birth
  Neonatal factors associated with executive functions disorders in former prematures in 3 to 4 year old and adequacy between BRIEF questionnaire performed/completed by parents and BRIEF questionnaire performed by teacher.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France

REFERENCES:
- [Derived] Reynold de Seresin M, Roy A, Theveniaut C, Le Goff J, Chopin C, Rouger V, Roze JC, Flamant C, Muller JB. Assessing of executive functions in daily life in preterm children aged 3-4 years old from the "Behavior Rating Inventory of Executive Function-Preschool version" questionnaire. Front Pediatr. 2023 Jul 26;11:999100. doi: 10.3389/fped.2023.999100. eCollection 2023. PMID 37565238